CLINICAL TRIAL: NCT02633475
Title: Association Between Interleukin-10 Promoter-1082A/G Polymorphism With Idiopathic Recurrent Miscarriage Risk of Chinese Han
Brief Title: Interleukin-10 Promoter-1082A/G Polymorphism and Idiopathic Recurrent Miscarriage Risk
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fourth Affiliated Hospital of Guangxi Medical University (Other)
Collaborators: Liuzhou Maternity and Child Healthcare Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PJK201583
Record Dates: First submitted 2015-12-11; First posted 2015-12-17 (Estimated); Last update posted 2017-02-15 (Actual); Status verified 2017-02

CONDITIONS: Abortion, Spontaneous
Keywords: interleukin-10; Polymorphism, Single Nucleotide
MeSH Terms: conditions — Abortion, Spontaneous

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — blood samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- CONTROL: women no miscarriage: Group of patients who referred to the Fourth Affiliated Hospital of Guangxi Medical University or Liuzhou Maternity and Child Healthcare Hospital, who have more than one successful pregnancy without miscarriage. Then the blood sample will be collected and the IL-10 Polymorphism will be analyzed.
  Interventions: Genetic: IL-10 polymorphism
- CASE: patients with IRM: Group of patients who referred to the Fourth Affiliated Hospital of Guangxi Medical University or Liuzhou Maternity and Child Healthcare Hospital, who have more than three consecutive miscarriages without clear cause (Idiopathic Recurrent Miscarriage, IRM). Then the blood sample will be collected and the IL-10 Polymorphism will be analyzed.
  Interventions: Genetic: IL-10 polymorphism

INTERVENTIONS:
Genetic: IL-10 polymorphism — The IL-10 genotype will determined by polymerase chain reaction (PCR) amplication and restriction length fragment polymorphisms.

SUMMARY:
This study aimed to assess the correlation between the interleukin-10 (IL-10)-1082A/G polymorphism and idiopathic recurrent miscarriage (IRM) of Chinese Han. A total of 100 women with IRM and 100 control women with a successful pregnancy will be included in this study. Then genotyping will be performed.

DETAILED DESCRIPTION:
As a common occurrence in early pregnancy, IRM has been associated with multiple causes, among which the disorders of immune homeostasis between the fetus and the maternal immune system, maintained by cytokines from the complex regulatory network, are considered one of the potential etiological factors underlying IRM.

The IL-10 polymorphism -1082A/G (rs1800896), which is located in the promoter region of the IL-10 gene, was reported to be implicated in the abnormal expression of IL-10 in IRM by some studies.

However, no such reports about the association between IL-10 polymorphism -1082A/G and IRM risk in Chinese Han.

ELIGIBILITY:
Inclusion Criteria:

1. women with more than three consecutive unexplained pregnancy losses before the 20th week;
2. Chinese Han Population;
3. Patients who signed informed consent.

Exclusion Criteria:

1. Patients who had other high-risk factors which might relate with recurrent miscarriage, including: (1) Parental karyotype abnormalities: significant rearrangements (e.g. balanced translocations and mosaics) were considered abnormal. If either the patient (or her partner) had an abnormal karyotype, it was considered a parental karyotypic abnormality; (2) Genital tract abnormalities: Any congenital anatomical deformation of the genital tract was considered abnormal; intrauterine adhesions, endometriosis and hydrosalpinx were also considered abnormal; (3) alloimmune disorder; (4) Endocrine abnormalities: prolactin (PRL) level >25 ng/ml, testosterone level >2.6 nmol/L, thyroid-stimulating hormone level <0.30 mU/L or >4.5 mU/L, free thyroxine (FT4) level <8.36 nmol/L or >29.6 nmol/L and free triiodothyronine (FT3) level <1.84 nmol/L or >7.39 nmol/L. Glucose level > 126mg/dl; (5) Autoimmune disorders: Any positive results of Anti-cardiolipin antibodies (ACA-IgG/IgM/IgA), anti-nuclear antibodies (ANA-IgG), anti-endometrium antibodies (AEA-IgM), anti-ovary antibodies (AOA-IgM), anti-sperm antibodies (ASA-IgM), antithyroidin(TG-Ab), anti-thyroid peroxidase antibody(TPO-Ab) and/or anti-chorionic gonadotropin hormone antibody; (6) Hypercoagulation state: D-dimer levels >260 ng/ml, fibrin degradation products (FDP) levels >5 mg/L or anti-beta 2-glycoprotein I (anti-beta 2-GP1) levels >15 U/ml; (7) Negative RH blood groups; (8) Abnormal semen routine results of patients husband.
2. Patients with serious diseases;
3. Patients with administration of contraceptive pills;
4. Patients participated in other randomized clinical research;
5. Patients could not be followed-up of a long time or had poor compliance;
6. Patients with other factors that would affect the study result.

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Female patients who referred to the Fourth Affiliated Hospital of Guangxi Medical University or Liuzhou Maternity and Child Healthcare Hospital
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2015-08; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
genetic polymorphisms associated with idiopathic recurrent miscarriage | within one year (plus or minus 1 month) after surgery
  Identification of genetic polymorphisms that are associated with idiopathic recurrent miscarriage

SECONDARY OUTCOMES:
Indexes in the routine blood test and blood coagulation test | During pregnancy and three months after miscarriage
  To explore the differential indexes in the routine blood test and blood coagulation test between patients with idiopathic recurrent miscarriage and healthy women, such as: WBC, NEU, LYM, RBC, HB, RDW, MCV, PLT, MPV, PDW, PCT, Fib, D-dimer.

CONTACTS AND LOCATIONS:
Overall Officials: Xiangcheng Wei, Principal Investigator — Guangxi Medical University Institutional Review Board
Locations (2):
- China (2):
  - Liuzhou Maternal and Child Health Care Hospital, Liuchow, Guangxi
  - the Fourth Affiliated Hospital of Guangxi Medical University, Liuchow, Guangxi

IPD SHARING:
Plan to Share IPD: No